CLINICAL TRIAL: NCT07362381
Title: A Randomized Controlled Trial to Address a Multimodal Intervention in the Elderly: the Efficacy of the CAMINN Study
Brief Title: A Randomized Controlled Trial to Address a Multimodal Intervention in the Elderly
Acronym: CAMINN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Collaborators: Ingesan-OHLA (Unknown)
Responsible Party: Principal Investigator, Guillermo Palacios, Associate Professor, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Protocol 3243/2023
Record Dates: First submitted 2026-01-05; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: People 60 Years of Age or Over 55 Years of Age With a Diagnosed Pathology and Preferably With a Recognized Physical and/or Cognitive Dependency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group receives treatment
  Interventions: Other: Multimodal intervention in the elderly
- Control (No Intervention): Control group

INTERVENTIONS:
Other: Multimodal intervention in the elderly — To measure the effectiveness of the intervention, eight variables were assessed: cognitive impairment, quality of life, depression, perceived loneliness, functional capacity to perform basic activities and tasks of daily living (ADL), ability to perform instrumental activities of daily living (iADL) and balance and gait. The following inventories were used as instruments to measure the aforementioned variables at baseline, mid intervention and after intervention: MMSE scale, FUMAT scale, the abbreviated version of the Yesavage Geriatric Depression Scale, the revised ESTE scale, the Barthel's scale, the Lawton and Brody's test and the Tineti's scale.
  Arms: Experimental group

SUMMARY:
The study is a quantitative randomized control trial (RCT) with a longitudinal pre-test, mid-test and post-test within and between subject design. It was conducted between July 2023 and December 2024. This study has been developed under a multicenter basis, since the intervention has involved institutionalized participants in two different nursing homes/care facilities as well as participants in community-dwelling settings. Participants were randomly allocated to two groups (experimental and control). Randomization was performed by means of a computer-generated random number schedule. The trial began with 187 participants. The objective of the intervention was to determine if after the application of a multimodal intervention for 18 months, the subjects would obtain significant improvements in the scores of different clinically validated tests

ELIGIBILITY:
Inclusion Criteria:

* be over 60 years of age or over 55 years of age with a diagnosed pathology and preferably with a recognized physical and/or cognitive dependency; have the cognitive capacity to maintain fluid conversations and repeat movements through a video call with a professional; be able to acquire the ability to connect autonomously to sessions or have a reference person in charge of the connections; the person must have a television with an HDMI input port.

Exclusion Criteria:

* severe cognitive impairment, situations of great physical dependence that lack help, or psychotropic substance abuse or dependence.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
quality of life | up to 18 months
  The FUMAT scale (Gómez et al., 2008) was used to assess quality of life by means of 8 different dimensions. The higher the score across its eight dimensions, the greater the individual's perceived and objective quality of life. It assesses areas such as emotional well-being, relationships, material well-being, personal well-being, physical well-being, self-determination, inclusion, and rights.
  Gómez, L. E., M. A., V., Arias, B., & Navas, P. (2008). Evaluación de la calidad de vida en personas mayores y con discapacidad: La Escala Fumat. Intervención Psicosocial, 17(2). https://doi.org/10.4321/S1132-05592008000200007
Cognitive impairment | up to 18 months
  Cognitive impairment was assessed via the Mini Mental State Examination, MMSE) (Folstein et al., 1975). The MMSE (Mini-Mental State Examination) is a 5-10 minute screening test that assesses cognitive status (orientation, memory, attention, language) through 30 simple questions and tasks. It is scored out of 30, where 24 points suggest cognitive impairment. A higher score indicates better cognitive function.
  Folstein, M. F., Folstein, S. E., & McHugh, P. R. (1975). "Mini-mental state." Journal of Psychiatric Research, 12(3), 189-198. https://doi.org/10.1016/0022-3956(75)90026-6
depression | up to 18 months
  The abbreviated version of the Yesavage Geriatric Depression Scale (Martínez de la Iglesia et al., 2002) was used to assess depression.
  The 15-item Abbreviated Geriatric Depression Scale (GDS-15), validated in Spanish by Martínez de la Iglesia et al. (2002), is a reliable, Yes/No questionnaire used to screen for depression in adults over 65. It offers similar diagnostic accuracy to the original 30-item version, typically using a cutoff score >= 5 to indicate depression
perceived loneliness | up to 18 months
  Loneliness was assessed using the revised ESTE scale (ESTE-R) (Rubio & Aleixandre, 1999). The ESTE scale is a psychometric tool designed to measure unwanted loneliness in older adults, assessing three key factors: social support, use of new technologies, and social participation. It uses a questionnaire that scores from 0 to 30, determining low, medium, or high levels of loneliness. The higher the total score, the greater the level of loneliness reported by the individual.
  Rubio, R., & Aleixandre, M. (1999). La escala "Este", un indicador objetivo de soledad en la tercera edad. Geriatrika. Revista Iberoamericana de Geriatría y Gerontología, 15, 26-35.
Activities of daily living (ADL) | up to 18 months
  The Barthel's scale (F.I. Mahoney & Barthel, 1965) was used to measure the subjects' functional capacity to perform basic activities and tasks of daily living (ADL).The Barthel's scale is a functional assessment tool that measures a person's independence in 10 basic activities of daily living (ADLs) using a score from 0 to 100. It is based on observation or questioning about the ability to eat, bathe, dress, control bowel and bladder control, transfer, and ambulate. A higher score on the scale indicates a greater level of independence.
  F.I. Mahoney, & Barthel, D. W. (1965). Functional Evaluation: The Barthel Index. Md State Med J., 14, 61-65.
Instrumental activities of daily living (iADL) | up to 18 months
  Lawton and Brody's test (Lawton & Brody, 1970) was used to measure the ability to perform instrumental activities of daily living (IADL). The Lawton and Brody Scale is a geriatric tool that measures the independence of older adults in performing Instrumental Activities of Daily Living (IADLs). It assesses eight key areas, such as using the telephone, shopping, preparing food, household chores, laundry, transportation, medication management, and finances. Scores are assigned from 0 (dependent) to 1 (independent) per item, for a total of 0 to 8, indicating the degree of autonomy and allowing for early detection of functional decline. Higher scores on the scale indicate greater independence.
  Lawton, M. P., & Brody, E. M. (1970). Assessment of older people: Self-maintaining and instrumental activities of daily living. Nursing Research, 13(3), 278.
Tinetti scale | up to 18 months
  Tineti's scale (Tinetti, 1986) was used to assess the balance and gait of older adults and determine the risk of falls. The Tinetti scale is a geriatric assessment tool that measures the risk of falls in older adults by analyzing their balance and gait through direct observation. It scores everyday tasks (sitting, standing, turning, walking) on a scale of 0 to 28, where less than 19 points indicates high risk and more than 25 indicates low risk.
  Tinetti, M. E. (1986). Performance-oriented assessment of mobility problems in elderly patients. J Am Geriatr Soc., 34, 119-126.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zaragoza, Teruel, Teruel, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2026-01-14): https://cdn.clinicaltrials.gov/large-docs/81/NCT07362381/Prot_SAP_000.pdf